CLINICAL TRIAL: NCT03323060
Title: A Multicenter Post-Market Clinical Follow-Up of the Medrobotics Flex Robotic System and Flex Rectoscope Used for Accessing and Visualizing the Anus, Rectum, and Distal Colon During Transanal Procedures
Brief Title: Post-Market Clinical Follow-Up to Access & Visualize the Anus, Rectum, & Distal Colon During Transanal Procedures
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medrobotics Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: FLX-CRC-PMK-US-001
Record Dates: First submitted 2017-10-20; First posted 2017-10-26 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Disease or Lesions of the Anus, Rectum, or Distal Colon
MeSH Terms: conditions — Disease | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Male and/or females ≥ 22 yrs old: ≥ 22 years of age requiring transanal procedures in the areas of the anus, rectum, and distal colon Transanal endoscopic surgical procedure
  Interventions: Device: Transanal endoscopic surgical procedure

INTERVENTIONS:
Device: Transanal endoscopic surgical procedure — Resection of tumors or lesions
  Other Names: Laparoscopy

SUMMARY:
To assess the safety and performance of the Medrobotics Flex Robotic System and Flex Rectoscope for accessing and visualizing the Anus, Rectum, and Distal Colon when used for Transanal procedures

ELIGIBILITY:
Inclusion Criteria:

* ≥ 22 years of age
* Candidate for transanal procedures in the areas of the anus, rectum, and distal colon.

Exclusion Criteria:

* Candidates are excluded if they < 22 years of age and do not meet criteria for transanal surgery in the anus, rectum, and distal colon

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 22 years of age requiring transanal procedures in the areas of the anus, rectum, and distal colon
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Access and Visualization | 0-24 hours
  Ability to access/touch with compatible flexible instruments and visualize/see with the scope/camera each of the four anatomical locations in the anus, rectum, and distal colon. The 4 areas to be accessed/touched and visualized/seen from the most proximal to the most distal are; Lower Rectum, Mid Rectum, Upper Rectum, Rectosigmoid Junction

SECONDARY OUTCOMES:
Performance of transanal surgical procedure | 0-24 hours
  Ability to complete the planned transanal surgical procedure using the Flex Robotic System, Flex Rectoscope and Flex compatible flexible instruments

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Univsersity of Nevada School of Medicine, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York